CLINICAL TRIAL: NCT05832476
Title: O-GlcNac Modified Proteomics Study of the Maturation of Hemodialysis Arteriovenous
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201712231RINC
Record Dates: First submitted 2023-04-14; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2018-01

CONDITIONS: Arteriovenous Fistula Occlusion
Keywords: Arteriovenous Fistula; vascular smooth muscle; histological technique; O-GlcNac; proteomics
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Matured: It is defined as the target HDAVF can be used
  Interventions: Other: No intervention
- Non-matured: RC-AVF underwent additional intervention after 90 days of observation
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
We divided into three parts to carry out. Firstly, evidence the pre-existing fibrosis in vein of AVF failure patients. investigation of expression, the role, and the mechanism by which the identified O-GlcNAac proteins promote, maturation of AV fistula. Finally, ddress and compare the proteomics differentiation between failure and maturation of AVF patients.

DETAILED DESCRIPTION:
End stage renal disease (ESRD) patients requires hemodialysis to maintain bloodstream functions. Before the hemodialysis, the patients requires a long-term vascular access, which best choice is Arteriovenous fistulas (AVF). However, 1/3 of patients were failure in AVF maturation, and it is still unknown. Our preliminary data have shown that pre-exisiting fibrosis in vein of AVF failure. Here, we will investigate whether pre-existing fibrosis of vein is asssociated with circulating fibrocytes in AVF failure, and further to address molecular mechanism of fibrocytes differentiation. We will divide into three parts to carry out. Firstly, evidence the pre-existing fibrosis in vein of AVF failure patients. Secondary, investigation of expression, the role, and the mechanism by which the identified O-GlcNAac proteins promote, maturation of AV fistula. Finally, address and compare the proteomics differentiation between failure and maturation of AVF patients. We hope that through this project, we can obtain signifiture molecules for precision detection and solve the current clinical unmet need.

ELIGIBILITY:
Inclusion Criteria:

* Age of 20 and older adult patients, and preoperatively clinical and ultrasound assessment of the arm vessels are fisible for the creation of a native HDAVF that include:the augmented diameters of the veins is > 2.0 mm and the diameter of the radial artery is> 2.0 mm. Besides, there is no obvious stenosis of vessels in the forearm.

Exclusion Criteria:

* The patient refused to join the study
* Too weak
* Serious heart failure
* Unconsciousness
* Bedridden for long time
* systemic lupus erythematosus(SLE), or other known autoimmune diseases
* The physician excludes the possibility of creating a wrist HDAVF before surgery
* Surgeon preoperatively identifies vessel inadequacy for the creation of a wrist HDAVF
* Choose a site other than the wrist for surgery
* Unexpected negative complications happen during surgery that prevent the completion of a wirst HDAVF

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age of 20 and older adult patients, and preoperatively clinical and ultrasound assessment of the arm vessels are fisible for the creation of a native HDAVF that include:the augmented diameters of the veins is > 2.0 mm and the diameter of the radial artery is> 2.0 mm. Besides, there is no obvious stenosis of vessels in the forearm.
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-10-26 (Actual)

PRIMARY OUTCOMES:
The diameter of each passage of the passage vein (forearm head vein) of the arterial and venous access within three months | Postoperative Three months
  Comparison of the various methods to achieve within three months the checkpoint path diameter increase rate (two time points measurement difference).

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Yang Chan, phd, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, No.7, Chung Shan S. Rd, Taiwan

IPD SHARING:
Plan to Share IPD: Yes